CLINICAL TRIAL: NCT04006821
Title: PD-1 Antibody Combined With Apatinib Mesylate as 2+ Line Treatment of Serum AFP-elevated Gastric Adenocarcinoma: an Open-label, Single-arm, Multicenter Phase II Study
Brief Title: PD-1 Antibody + Apatinib Mesylate in 2+ Line Serum AFP-elevated Gastric Adenocarcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Medical University, China (Other)
Responsible Party: Principal Investigator, Jingdong Zhang, Director, China Medical University, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PD-1-APTN-Ⅱ-AFPGC
Record Dates: First submitted 2019-07-01; First posted 2019-07-05 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Gastric Cancer; AFP
MeSH Terms: conditions — Stomach Neoplasms | interventions — spartalizumab; camrelizumab; apatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PD-1 antibody + Apatinib mesylate (Experimental): Every patient will receive PD-1 antibody 200mg iv every 2 weeks and apatinib 250mg or 500mg (according to the patient's tolerance) orally every day. PD-1 antibody will be administered until disease progression or lasts for two years. Apatinib mesylate will be administered until disease progression.
  Interventions: Drug: PD-1 antibody; Drug: Apatinib mesylate

INTERVENTIONS:
Drug: PD-1 antibody — Camrelizumab will be administered 200mg iv every 2 weeks until disease progression or lasts for two years.
  Other Names: Camrelizumab
Drug: Apatinib mesylate — Apatinib mesylate will be administered 250mg or 500mg (according to the patient's tolerance), qd, oral, until disease progression.

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of PD-1 antibody combined with apatinib mesylate in patients with unresectable, local advanced recurrent or metastatic serum AFP-elevated gastric adenocarcinoma, who have at least received first-line antitumor therapy or whose standard treatment is intolerable.

DETAILED DESCRIPTION:
AFP-elevated gastric adenocarcinoma is a special type of gastric cancer, with the characteristics of high risk of liver and lymph node metastasis, poor therapeutic effect, and prognosis.

This prospective study is a single-arm, open-label, multi-center phase II clinical trial to evaluate the efficacy and safety of PD-1 antibody combined with apatinib mesylate in patients with unresectable, local advanced recurrent or metastatic serum AFP-elevated gastric adenocarcinoma, who have at least received first-line antitumor therapy or whose standard treatment is intolerable.

AFP elevation is defined as serum AFP > 20 ng/ml. In this prospective study, the objective remission rate (ORR) will be used as primary outcome measures and 30 patients will be recruited. PD-1 antibody combined with apatinib mesylate will be administered. PD-L1 expression and TMB will be measured before treatment. In addition, the dynamic changes of serum AFP levels, T lymphocyte in peripheral blood will be monitored before each treatment cycle. In the course of treatment, safety evaluation will be carried out according to the standard of adverse reaction classification (CTCAE) 4.0.

ELIGIBILITY:
Inclusion Criteria:

* Patients must volunteer to participate in the study, signed informed consent, and were able to comply with the program requirements of visits and related procedures.
* Age and gender: ≥18 years old and≤75 years old, both men and women.
* All subjects must have unresectable, local advanced recurrent or metastatic gastric cancer, and have histologically confirmed predominant adenocarcinoma with serum AFP-elevated (serum AFP > 20 ng/ml).
* Subject must have at least received first-line antitumor therapy or whose standard treatment is intolerable.
* Subject must have at least one measurable lesion or evaluable disease by CT or MRI per iRECIST 1.1 criteria.
* Subject must be previously untreated with anti-angiogenesis molecular targeted therapy and immunotherapy for gastric cancer (including anti-CTLA-4, PD-1/PD-L1 monoclonal antibody immunotherapy).
* ECOG performance status score of 0 or 1.
* Child-Pugh score < 6 (Child-Pugh A), and no history of hepatic encephalopathy.
* Expected survival: ≥12 weeks.
* Adequate bone marrow, hepatic and renal function as assessed by the following laboratory requirements conducted within 7 days of starting study treatment:

Neutrophil count≥1.5×10^9/L; Platelet count≥80×10^9/L; Hemoglobin≥90g/L; Serum albumin≥28g/L; Total bilirubin (TBI)≤1.5×ULN; Alanine aminotransferase (ALT)≤3×ULN (or≤5×ULN if liver metastases are present); Aspartate aminotransferase (AST)≤1.5×ULN (or≤5×ULN if liver metastases are present); Alkaline phosphatase (ALP)≤2.5×ULN Thyrotropin (TSH) ≤1×ULN (FT3 and FT4 levels should be examined at the same time if abnormal, such as FT3 and FT4 levels are normal, can be included in the group); Serum creatinine≤1.5×ULN or calculated creatinine clearance≥40 mL/min (using the Cockcroft-Gault formula) Female CrCl = (140- age in years) × weight in kg × 0.85 / 72 × serum creatinine in mg/ dL Male CrCl = (140- age in years) × weight in kg × 1.00 / 72 × serum creatinine in mg/ dL Subjects not receiving anticoagulation therapy: INR or APTT ≤ 2×ULN; Urine protein < 2+; 24-hour urinary protein content <1.0g/24-hour if urinary protein ≥2+;

* Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test within 72 hours prior to the start of study drug. WOCBP must agree to follow instructions for method(s) of contraception (e.g. intrauterine devices, contraceptives or condoms) for the duration of study treatment and 3 months after the last dose of study treatment. Subjects must be non-lactating. Males who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of study treatment and 3 months after the last dose of study treatment.
* If HBsAg (+) and/or HBcAb (+), HBV DNA is required to be <500 IU/mL, and the original anti-HBV treatment is continued throughout the study period, or start to anti-HBV treatment throughout the study.

Exclusion Criteria:

* With history of active autoimmune disease or autoimmune disease (For example, the following, but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, pituitary, vasculitis, nephritis, hyperthyroidism; patients with vitiligo; in childhood asthma has been completely alleviated, adults without any intervention can be included; asthma with medical intervention could not be included). Substitution therapy is not considered as systemic therapy. Patients with the following diseases are not excluded and may proceed to further screening:

  1. Controlled Type I diabetes
  2. Hypothyroidism (provided it is managed with hormone replacement therapy only)
* Any condition that required systemic treatment with either corticosteroids (> 10 mg daily of prednisone or equivalent) or other immunosuppressive medication ≤ 14 days before randomization.
* A history of severe allergy to any monoclonal antibody or anti-angiogenesis targeted drug.
* Patients with known central nervous system metastasis (suspected need to be excluded by MRI scans) or a history of hepatic encephalopathy.
* The total volume of liver metastases>50%, or obvious infiltration of bile duct or portal vein trunk, or patients who have received liver transplantation in the past.
* More than a small amount of pericardial effusion, uncontrollable pleural effusion or ascites requiring frequent drainage or medical intervention.
* Uncontrollable hypertension with drugs (systolic pressure ≥140 mmHg or diastolic pressure≥90 mmHg).
* With history of serious cardiovascular and cerebrovascular diseases:

Any history of heart failure meeting New York Heart Association Classification III or IV ≤3 months before randomization； Left ventricular ejection fraction < 50% by color Doppler echocardiography； Uncontrolled arrhythmias or unstable angina pectoris； Corrected QT interval > 500ms (calculated by Fridericia method).

* Abnormal coagulation function (INR > 2.0, PT > 16s), with haemorrhagic tendency or undergoing thrombolytic or anticoagulant therapy, but prophylactic use of low-dose aspirin and low-molecular-weight heparin is allowed.
* Significant clinical bleeding symptoms or definite bleeding tendency occurred within 3 months before randomization.
* Arteriovenous thrombosis events occurring within 6 months before randomization.
* Hereditary or Acquired Hemorrhage and Thrombosis Tendency.
* Metastatic diseases involving major airways or blood vessels or large central mediastinal tumors.
* Urinary routine indicated that urinary protein (++) and confirmed 24-hour urinary protein content > 1.0 g.
* Has received any radiotherapy, chemotherapy, hormone therapy, surgery or any investigational therapies within 28 days or 5 half-lives (whichever is longer) of the first study drug administration.
* Patients with toxicities (as a result of prior anticancer therapy) which have not recovered to baseline or ≤ CTCAE 1, except for AEs not considered a likely safety risk (eg, alopecia and specific laboratory abnormalities).
* Systemic immunostimulants (including interferon and IL-2) were administered within 28 days or 5 half-lives (whichever is longer) before randomization. Systemic immunosuppressive drugs (such as glucocorticoids) were administered within 2 weeks, or systemic immunosuppressive drugs were expected to be used during the study period. Patients who are currently or have previously been on any of the following steroid regimens are not excluded:

Acute, low-dose systemic immunosuppressive drugs or single-shot systemic immunosuppressive drugs (e.g. 48-hour glucocorticoid administration to prevent and treat contrast agent allergy); Treatment of chronic obstructive pulmonary disease or bronchial asthma with corticosteroids inhalation administration such as fluorocortisone and glucocorticoids; Accept low doses of glucocorticoid to treat postural hypotension or adrenal insufficiency (dose ≤ 10 mg daily of prednisone or equivalent).

* With severe chronic or active infections (including tuberculosis infection, etc.) requiring systemic antibacterial, antifungal or antiviral therapy within 7 days of the first study drug administration.
* Abdominal or tracheoesophageal fistula, gastrointestinal (GI) perforation, intraperitoneal abscess or intestinal obstruction occurred within 6 months before randomization. Subjects with incomplete obstructive/obstructive syndrome/intestinal obstructive symptoms/signs who have undergone definite surgical treatment and whose symptoms disappear are not excluded.
* Major surgical procedures (craniotomy, thoracotomy or laparotomy, etc.), open biopsy or major trauma, abdominal surgery or major abdominal trauma within 60 days prior to the start of treatment, or anticipated need for major surgical procedures during the study period, and not recovered from side effects. Tissue (hollow needle) biopsy or other minor surgery was performed within 3 days before randomization, except for the placement of intravenous infusion system devices.
* Congenital or acquired immunodeficiency (e.g. HIV-infected persons).
* Any active malignancy ≤ 5 years before randomization except for the specific cancer under investigation in this study and any cured limited tumors (eg, carcinoma in situ of the cervix or prostate, basal cell skin cancer).
* With history of interstitial lung disease, non-infectious pneumonitis.
* Gastric surgery and/or local treatment or experimental drug therapy for gastric cancer were performed within 4 weeks before randomization. In patients with bone metastasis, palliative radiotherapy for bone metastasis lesions within 1 week before randomization can be included (but the radiotherapy area is required to be less than 5% of the bone marrow area).
* Received prior therapies targeting PD-1, PD-L1, or PD-L2, or Apatinib mesylate.
* Was administered a live vaccine ≤ 4 weeks before randomization; or plan to live vaccinate during against PD-1 monoclonal antibody treatment or within five months after last administration.
* Concurrent participation in another therapeutic clinical trial, unless participating in observational (non-interventional) clinical studies or at the follow-up stage of interventional studies.
* Other situations that the researchers think should be excluded.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-07-25 (Actual); Primary Completion 2022-08-01 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 2 years
  The proportion of patients whose best overall response (BOR) is complete response (CR) or partial response (PR) assessed by iRECIST v1.1

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 2 years
  The time from the date of randomization to the date of first documentation of disease progression or death, whichever occurs first
Overall survival (OS) | 2 years
  The time from the date of randomization until the date of death due to any cause
6-month/9-month/12-month survival rate | 6-month/9-month/12-month
  After date of randomization, evaluate patient survival rate at 6,9 and 12 months, respectively.
Duration of response (DOR) | 2 years
  The time from complete response (CR) or partial response (PR) to disease progression or death
Disease control rate (DCR) | 2 years
  The proportion of patients whose BOR is CR, PR, and stable disease (SD) assessed
Incidence of Treatment-Emergent Adverse Events | 2 years
  The grade of toxicity will be assessed using the NCI-CTCAE version 4.0
Quality of life (QLQ C30) | Every 2 weeks after the first treatment until 2 years
  Scores according to EORTC QLQ-C30 scoring manual
Exploration of biomarkers | 2 years
  PD-L1 expression, TMB, changes of AFP and T lymphocyte in peripheral blood，and etc

CONTACTS AND LOCATIONS:
Overall Officials: Jingdong Zhang, Principal Investigator — China Medical University, China
Locations (1):
- Cancer Hospital of China Medical University/Liaoning Cancer Hospital &Institute, Shenyang, Liaoning, China